CLINICAL TRIAL: NCT02078206
Title: Early Neurocognitive Rehabilitation in Intensive Care
Acronym: ENRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Lluis Blanch, PhD, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPT-2013/057
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness
Keywords: Critical illness; Neurocognition; Neurocognitive stimulation; Delirium; Virtual Reality; cognitive; rehabilitation; ICU
MeSH Terms: conditions — Critical Illness; Delirium

ARMS (2):
- Neurocognitive stimulation (Experimental): Intervention of experimental group consists in a neurocognitive stimulation treatment. Using kinect technology, patient can interact with a virtual environment where different cognitive tasks have to be resolved.
  Interventions: Other: Neurocognitive stimulation
- Treatment as usual (No Intervention)

INTERVENTIONS:
Other: Neurocognitive stimulation
  Arms: Neurocognitive stimulation

SUMMARY:
The purpose of this project is to assess the efficacy of an early neurocognitive intervention for ICU patients, in terms of psychopathological, neuropsychological and functional improvement. The treatment is supported in an interactive advanced computing platform that includes the continuous biomedical registration of the patients and a virtual reality software specifically designed for critical patients.

The investigators expect an improvement in neuropsychological, psychopathological and functional status at hospital discharge and 3 months follow-up in those patients that have received the early neurocognitive intervention comparing with patients treated as usual. Furthermore the investigators expect a decrease of episodes and/or duration of delirium in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years
* Patients receiving mechanical ventilation for at least 24 hours
* Patients scoring more than 8 on the Glasgow Coma Scale (GCS) and more than 2 on the Sedation Agitation Scale (SAS)
* Patients haemodynamically stable
* Informed consent signed by the closest relatives.

Exclusion Criteria:

* Patients with previous neurologic pathology or focal brain injury before ICU admission
* Patients with serious psychiatric pathology (major depression, psychosis, bipolar disease) or mentally retarded
* Patients with sensorial alterations needed to interact with the neurocognitive stimulation programme
* patients whose closest relatives refuse the subject to be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Attention | Hospital discharge and 3-months after hospital discharge
  * Verbal attention: Digits Forward subtest of the WAIS III (Wechsler, 1999)
  * Visual attention: Spatial Localization Forward subtest of the WMS III (Wechsler, 1999)
  * Sustained/Selective attention: Continuous Performance Test (Conners, 1992)
Memory | Hospital discharge and 3-months after hospital disharge
  * Verbal learning and memory: Auditory Verbal Learning Test (Rey, 1964)
  * Visual learning and memory: 10/36 Spatial Recall Test (Rao, 1992)
  * Visual recognition: Benton Visual Retention Test (Benton, 1983)
Executive Functions | Hospital discharge and 3-months after hospital discharge
  * Stimuli alternation and sequencing: Trail Making Test A-B (Mimeo & Manga, 1999)
  * Automatic inhibition response: Stroop Test (Golden & Charles, 1978)
  * Visual planning: Tower of London (Shallice, 1982).
  * Phonetic verbal fluency: FAS test (Spreen and Benton, 1995)
  * Semantic verbal fluency: Animals 1' (Benton & Hamsher, 1976)
Speed processing | Hospital discharge and 3-months after hospital discharge
  - Information processing speed: Symbol Search subtest of the WAIS III (Wechsler, 1999)
Psychopathological status | Hospital discharge and 3-monts after hospital discharge
  * Depression: Hamilton Depression Rating Scale (HDRS) (Hamilton, 1960)
  * Anxiety: Hamilton Anxiety Rating Scale (HAM-A) (Hamilton, 1959)
Functional Status | hospital discharge and 3-months after hospital discharge
  * Quality of life questionnaire: Satisfaction and Pleasure (Q-LES-Q) (Endicott, J., Nee, J., Harrison, W. & Blumenthal, R., 1993)
  * Lawton and Brody Functional Scale (1969)

SECONDARY OUTCOMES:
Delirium | Every day during ICU stay
  Number of episodes and duration of delirium: Confusional Assessment Method for Intensive Care Unit (CAM-ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Blanch, Phd, Principal Investigator — Fundació Parc Taulí; Antoni Artigas, Phd, Study Director — Corporació Parc Taulí- Critical Care Unit chair
Locations (1):
- Corporació Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Turon M, Fernandez-Gonzalo S, Jodar M, Goma G, Montanya J, Hernando D, Bailon R, de Haro C, Gomez-Simon V, Lopez-Aguilar J, Magrans R, Martinez-Perez M, Oliva JC, Blanch L. Feasibility and safety of virtual-reality-based early neurocognitive stimulation in critically ill patients. Ann Intensive Care. 2017 Dec;7(1):81. doi: 10.1186/s13613-017-0303-4. Epub 2017 Aug 2. PMID 28770543